CLINICAL TRIAL: NCT00241566
Title: Economic Medical Evaluation of Treatment of the Neuropathic Pain Rebel by Cortical Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pr Jean-Jacques LEMAIRE, CHU Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0002
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Neuropathic Pain Rebel
Keywords: Neuropathic pain; Electric cortical stimulation; Economic Medical evaluation
MeSH Terms: conditions — Neuralgia

INTERVENTIONS:
Device: implantation of stimulator

SUMMARY:
All neuropathic chronicle pains are difficult to treat. Currently many patients are not relieved by electric stimulations of central nervous system, existing. Recently cortical stimulation had a development important and benefit effects are proven. In this study we evaluate medico-economic impact of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of pain caused by lesion of central or peripheral nervous system
* Pain persistent since one year at least
* Pain untreated with 3 different antalgic treatments

Exclusion Criteria

* Pain linked t a malignant affection
* patient < 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-08; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cost of treatment of this pathology

SECONDARY OUTCOMES:
Evaluation of the pain when the electric stimulation is off or on (during one month for each one). Using Visual Analogic Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Lemaire, Principal Investigator — Clermont-Ferrand UH
Locations (2):
- France (2):
  - Clermont-Ferrand UH, Clermont-Ferrand, Auvergne
  - Neurosurgery - Henri Mondor Hospital, Créteil, Île-de-France Region